CLINICAL TRIAL: NCT05321771
Title: The Effect of Involving a Family Caregiver in Promoting the Principles of the Hospital Elder Life Program on Decreasing Delirium Among Older Patients Hospitalized in the Orthopedic Unit Following Surgery for Post-fall Femoral Fracture.
Brief Title: Family Caregiver Role in Decreasing Delirium in Older Patients With Fractured Femur Using HELP Principles.
Acronym: FamHelp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Tzvi Dwolatzky, Director Geriatrics, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0508-21-RMB
Record Dates: First submitted 2022-03-14; First posted 2022-04-11 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Delirium; Femoral Fracture
Keywords: Elderly; Acute hospitalization; Family caregiver; Hospital Elder Life Program
MeSH Terms: conditions — Delirium; Femoral Fractures

STUDY DESIGN:
Intervention Model Description: Single arm single center prospective interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family caregiver application of HELP principles (Experimental): The family caregiver will apply the principles of the HELP program in a structured manner following training by a nurse clinical specialist in geriatrics. The patient will be assessed daily by means of the Confusion Assessment Method (CAM) and the 4 'A's test (Arousal, Attention, Abbreviated Mental Test - 4, Acute change) (4AT) to determine delirium incidence.
  Interventions: Other: Family caregiver application of HELP principles

INTERVENTIONS:
Other: Family caregiver application of HELP principles — The family caregiver will apply the principles of the HELP program in a structured manner following training by a nurse clinical specialist in geriatrics. These principles include engaging patients in conversation, particularly emphasizing orientation to time and place, encouraging eating and drinking, and assisting with early mobility.

SUMMARY:
The Hospital Elder Life Program (HELP) has been shown to reduce delirium in hospitalized patients. In this study a family caregiver will apply the principles of the HELP program in a structured manner following training by a nurse clinical specialist in geriatrics. The effect of this intervention in decreasing delirium in older patients treated in an acute orthopedic unit for fractured femur following a fall will be evaluated.

DETAILED DESCRIPTION:
Approximately 30% of those aged 65 years and over will fall at least once a year. As many as 38% of all older people hospitalized following a fall are admitted with hip fractures and 93% of these will undergo surgical repair of the fracture (Ministry of Health, 2015). Fractured femur is associated with many complications. Delirium (acute confusional state) following surgery is one of the most common of these complications, it often results in adverse outcomes for both patients and caregivers (Tieges et al., 2021), and places great financial burden on the health system. It must be emphasized that delirium can be prevented, and when it occurs should be recognized and treated appropriately. The HELP (Hospital Elder Life Program) is an accepted evidence-based model that has been proven to be effective in reducing delirium at the time of acute hospitalization (Inouye et al., 1999). HELP (which has been implemented at the Rambam Healthcare Campus) is a volunteer-based program using non-pharmacological interventions that include engaging patients in conversation, particularly emphasizing orientation to time and place, encouraging eating and drinking, and assisting with early mobility (Inouye, 2000). The HELP program has been shown to reduce delirium by one-fifth in previous studies (Wang et al., 2020). In this study a family caregiver will apply the principles of the HELP program in a structured manner following training by a nurse clinical specialist in geriatrics. The effect of this intervention in decreasing delirium in older patients treated in an acute orthopedic unit for fractured femur following a fall will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 65 years and older
* Acute hospitalization in the orthopedic unit for fractured femur post-fall
* Expected or actual surgical intervention for treatment of fracture
* At least one family caregiver involved in supporting the patient during hospitalization

Exclusion Criteria:

* Documented conditions that have been clinically active during the previous 6 months: including psychiatric illness; cerebrovascular disease; brain malignancy; alcohol abuse; drug abuse
* Terminal disease
* Delirium
* Inability to assess for delirium due to advanced dementia or sensory deprivation (marked impairment of vision or hearing) or any other condition that limits communication with the patient

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium | From date of signing informed consent until the date of first documented diagnosis of delirium or hospital discharge, whichever came first, assessed up to a maximum of 100 days
  The incidence of delirium will be determined according to the results of patient assessment by means of the CAM and 4AT instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Galit Geller Bigelman, MA, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, North, Israel

IPD SHARING:
Plan to Share IPD: No
Data will be available to other researchers on request

REFERENCES:
- [Result] Tieges Z, Maclullich AMJ, Anand A, Brookes C, Cassarino M, O'connor M, Ryan D, Saller T, Arora RC, Chang Y, Agarwal K, Taffet G, Quinn T, Shenkin SD, Galvin R. Diagnostic accuracy of the 4AT for delirium detection in older adults: systematic review and meta-analysis. Age Ageing. 2021 May 5;50(3):733-743. doi: 10.1093/ageing/afaa224. PMID 33951145
- [Result] Inouye SK, Bogardus ST Jr, Charpentier PA, Leo-Summers L, Acampora D, Holford TR, Cooney LM Jr. A multicomponent intervention to prevent delirium in hospitalized older patients. N Engl J Med. 1999 Mar 4;340(9):669-76. doi: 10.1056/NEJM199903043400901. PMID 10053175
- [Result] Inouye SK, Bogardus ST Jr, Baker DI, Leo-Summers L, Cooney LM Jr. The Hospital Elder Life Program: a model of care to prevent cognitive and functional decline in older hospitalized patients. Hospital Elder Life Program. J Am Geriatr Soc. 2000 Dec;48(12):1697-706. doi: 10.1111/j.1532-5415.2000.tb03885.x. PMID 11129764
- [Result] Wang YY, Yue JR, Xie DM, Carter P, Li QL, Gartaganis SL, Chen J, Inouye SK. Effect of the Tailored, Family-Involved Hospital Elder Life Program on Postoperative Delirium and Function in Older Adults: A Randomized Clinical Trial. JAMA Intern Med. 2020 Jan 1;180(1):17-25. doi: 10.1001/jamainternmed.2019.4446. PMID 31633738